CLINICAL TRIAL: NCT04151316
Title: Study of Periodontal Tissues in Fixed Prostheses on Natural Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Enrico Gherlone, Head of Dental School, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: BOPT 1 unisr
Record Dates: First submitted 2019-09-30; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-09

CONDITIONS: Prosthetic Tissue Defect; Dental Prosthesis Complication; Dental Prosthesis Failure; Tissue Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vertical group (Experimental)
  Interventions: Procedure: crown preparation; Procedure: vertical preparation
- horizontal group (Experimental)
  Interventions: Procedure: crown preparation; Procedure: horizontal preparation

INTERVENTIONS:
Procedure: crown preparation — includes tooth preparation
Procedure: vertical preparation — type of vertical preparation on the tooth that accepts the crown
  Arms: vertical group
Procedure: horizontal preparation — type of horizontal preparation on the tooth that accepts the crown
  Arms: horizontal group

SUMMARY:
When the tooth is severely compromised, it needs a prosthetic crown. The tooth is prepared to allow the housing of the prosthetic crown without difficulty. This study aims to compare two different types of preparations to see with which of the two the gingival tissue reacts best.

ELIGIBILITY:
Inclusion Criteria:

1. Need for restoration by single-tooth prosthetic crown, due to destructive caries, coronal fracture, endodontically treated tooth, severe abrasion, aesthetic problems, remake of old incongruous prosthetic crown, other complications.
2. If there are incongruous conservative restorations (composite fillings or other materials) in the elements adjacent to the tooth to be treated, these must be restored before the prosthetic therapy and must not be modified during the protocol.
3. Absence of active periodontal disease
4. over the age of 18;
5. periodontal probing less than 4 mm in the tooth to be treated
6. absence of bleeding on probing
7. full-mouth plaque score (FMPS) and full-mouth bleeding scores (FMBS) < 20% at the start of the study
8. Patients according to protocol participation and informed consent signature.

Exclusion Criteria:

1. contraindication to dental treatment
2. active periodontal disease
3. systemic diseases that may affect periodontitis
4. Pregnant women
5. Patients in orthodontic therapy
6. inability to return to the controls or to follow oral hygiene maintenance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
variation of gingival thickness | 12 months
  Gingival thickness (GT) measured in millimetres in the mid-buccal area of the tooth, at the central point between the gingival margin and the gingival mucus junction (MGJ) using an endodontic specillus with a silicone stop put in contact with the soft tissue until the specillus reaches the hard surface. At the time of the initial measurement of the periodontal parameters, i.e.
variation of gingival thickness digital | The impression is taken before the final impression (t1), at 3 months (t2), 6 months (t3), 12 months (t4) and the 3D images are compared using software to evaluate the variation of the soft tissue.
  At the time of the initial measurement of the periodontal parameters, i.e. at the time 0 before the prosthetic preparation of the tooth element, a digital impression is taken in order to obtain a 3D image of the tissues around the tooth element to be rehabilitated.

SECONDARY OUTCOMES:
BOP | TO (before the therapy), T1 (1 month after placement of the temporary restoration), T2 (3 months after placement of the temporary restoration), T3 (6 months after placement of the temporary restoration), T4 (1 year after placement of the definitive)
  percentage of bleeding of the gingival sulcus of all dental elements using a millimeter periodontal probe
PPD | TO (before the therapy), T1 (1 month after placement of the temporary restoration), T2 (3 months after placement of the temporary restoration), T3 (6 months after placement of the temporary restoration), T4 (1 year after placement of the definitive)
  probing depth (PD), recorded in millimetres at 6 points for each tooth using a millimeter periodontal probe
Recessions | TO (before the therapy), T1 (1 month after placement of the temporary restoration), T2 (3 months after placement of the temporary restoration), T3 (6 months after placement of the temporary restoration), T4 (1 year after placement of the definitive)
  relative gingival recession (rREC), measured at 6 points for each tooth as the distance from the gingival margin (GM) to the apical edge of the acrylic template previously using a millimeter periodontal probe
aesthetic value | TO (before the therapy), T1 (1 month after placement of the temporary restoration), T2 (3 months after placement of the temporary restoration), T3 (6 months after placement of the temporary restoration), T4 (1 year after placement of the definitive)
  Aesthetic evaluation of soft tissue is performed with the Pink Aesthetic Score/White Aesthetic Score (PES/WES). The PES evaluation consists of 7 variables: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue texture and color.
  Mucosa is evaluated with WES, which consists of 5 variables: tooth shape, volume, color, surface texture, translucency/characterization.
  The mesial and distal papillas are measured for absence, completeness, incompleteness, while the other variables are measured by comparing them with the contralateral teeth in terms of vertical level (score of 2), small (≤1 mm) discrepancy (score of 1), or large (≥1 mm) discrepancy (score of 0). The maximum score will be 14 for PES and 10 for WES, which will mean a perfect match for soft tissue and hard tissue respectively.
patient's satisfaction: VAS scale | TO (before the therapy), T1 (1 month after placement of the temporary restoration), T2 (3 months after placement of the temporary restoration), T3 (6 months after placement of the temporary restoration), T4 (1 year after placement of the definitive).
  Patient satisfaction is analyzed by means of a VAS scale
Digital valuation of emergency profile | The angle of the emergence profile is evaluated first with the temporary (T0 first week) and then with the definitive(T1 after 3 month).
  The prosthetic contour is evaluated with the fingerprint to evaluate the angular width of the emergence profile.
  The amplitude of the angle evaluated is that formed between the emergence profile (part of the crown in contact with the soft tissues) and the long axis of the tooth.
  The angle of the emergence profile is evaluated by making a digital impression on the plaster model with the crowns inserted in the prosthetic abutment of the master model, first with the temporary and then with the definitive. The unit of measurement expressed by the digital instrument is always the same so it is a single measurement carried out in two different times.
Evaluation of the interproximal papilla | gap between the most coronal part of the papilla and the point of contact is measured and re-evaluated at 3 months (t2), 6 months (t3), 12 months (t4)
  Once the final crowns have been cemented, the distance between the point of contact and the interproximal papilla is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Giulia, Milan, Italy/MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
we'll set up electronic databases for each patient.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: in a year and a half, we'd produce the data and leave it available.